CLINICAL TRIAL: NCT03072316
Title: Case Control Study to Evaluate the Impact of Radiotherapy on Patients Undergoing DIEP Flap Breast Reconstruction
Brief Title: Impact of Radiotherapy on Patients Undergoing DIEP Flap Breast Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4283
Record Dates: First submitted 2015-04-13; First posted 2017-03-07 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; mastectomy; deep inferior perforator flap reconstruction; post mastectomy radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- SSM immediate DIEP: Unilateral skin sparing mastectomy with immediate DIEP
  Interventions: Other: 3D surface imaging; Other: semi-structured interview; Other: applanation tonometry
- SSM immediate DIEP and PMRT: Unilateral skin sparing mastectomy with immediate DIEP flap reconstruction and post mastectomy radiotherapy
  Interventions: Other: 3D surface imaging; Other: semi-structured interview; Other: applanation tonometry
- mastectomy, PMRT, delayed DIEP: simple mastectomy, post mastectomy radiotherapy adn then delayed DIEP reconstruction
  Interventions: Other: 3D surface imaging; Other: semi-structured interview; Other: applanation tonometry
- SSM, temporizing implant, PMRT then DIEP: Unilateral SSM with temporizing implant, PMRT and subsequent
  Interventions: Other: 3D surface imaging; Other: semi-structured interview; Other: applanation tonometry

INTERVENTIONS:
Other: 3D surface imaging — 3D photography
Other: semi-structured interview — qualitative analysis using semi structured interview
Other: applanation tonometry — measurement of breast compressibility

SUMMARY:
The investigators intend to undertake a study to investigate the effect of radiotherapy on deep inferior epigastric perforator flap reconstructions (DIEP). Adjuvant post-mastectomy radiotherapy (PMRT) is offered to women at high risk of chest wall recurrence. The perceived detrimental effect of radiotherapy on an immediate breast reconstruction and the "one-off" nature of autologous reconstruction leads some surgeons to recommend delayed reconstruction after mastectomy or to use a temporising implant with a view to planned exchange to autologous reconstruction after radiotherapy. However, there remains significant uncertainty in the literature about the impact of radiotherapy on autologous reconstructions. This study is a mixed methology study using patient reported outcome measures (PROMS), applanation tonometry (measure of breast compressibility), semi-structured interviews and 3 dimensional photography analysis to compare the aesthetic and impact on quality of life on the following groups of patients:

Patient groups:

1. Unilateral skin sparing mastectomy (SSM) with immediate DIEP flap reconstruction and PMRT (cases)
2. Unilateral SSM with immediate DIEP flap reconstruction and no PMRT (controls)
3. Unilateral simple mastectomy, PMRT, and subsequent delayed DIEP flap reconstruction (controls)
4. Unilateral SSM with temporizing implant, PMRT and subsequent conversion to DIEP (controls)

DETAILED DESCRIPTION:
Since 1997, breast cancer has been the most common cancer in the UK, accounting for 31% of all new cancers in women. According to the latest statistics published by Cancer Research UK, approximately 50,000 women were diagnosed with breast cancer in 2010(1). In the UK, 53% of women with symptomatic breast cancer and 27% of those with screen-detected breast cancer are treated surgically with mastectomy; therefore approximately 21,500 undergo a therapeutic mastectomy each year (2). Guidelines from the National Institute for Health and Clinical Excellence (NICE) recommend that immediate breast reconstruction is offered to women during the same operation as their mastectomy (3). The UK National Mastectomy and Breast Reconstruction Audit Second Report 2009 (4) states that 21% of their cohort underwent immediate breast reconstruction, thus one would expect approximately 4500 women to undergo immediate reconstruction each year in the UK.

A breast reconstruction should mimic the natural appearance of the breast in shape, volume and compliance, together giving a symmetrical result. Breast reconstruction ranges from implant-based methods to autologous free flap reconstruction, such as the deep inferior epigastric perforator (DIEP) flap, which was first popularised by Allen in 1994(5). In our unit, the DIEP flap has become one of the most reliable and popular methods of breast reconstruction, with flap failure rate of less than 1%. We, like others, view it as the current "gold standard" in breast reconstruction(6)(7)(8).

Adjuvant post-mastectomy radiotherapy (PMRT) is offered to women at high risk of chest wall recurrence. The perceived detrimental effect of radiotherapy on an immediate breast reconstruction and the "one-off" nature of autologous reconstruction leads some surgeons to recommend delayed reconstruction after mastectomy or to use a temporising implant with a view to planned exchange to autologous reconstruction after radiotherapy. However, there remains significant uncertainty in the literature about the impact of radiotherapy on autologous reconstructions . Initially, small case series supported the clinical bias that radiotherapy is detrimental to the autologous reconstruction but, more recently, larger series have challenged this view. Each study has flaws, such as being underpowered, having insufficient duration of follow up, not reporting patient satisfaction or not measuring volume objectively such that residual questions remain. A recent systematic review by Kelley et al attempted to address questions related to complications and flap compromise as a result of radiation delivery before or after autologous breast reconstruction. The review analysed 20 articles with over 1,500 flap reconstructions. No significant differences in measurable postoperative complications including total flap loss, wound healing complications, infection, haematoma, seroma, and fat necrosis were found in comparing patients who underwent PMRT before or after autologous reconstruction. However, differences in cosmetic outcome and patient satisfaction in the irradiated and unirradiated flap reconstruction groups were not adequately addressed.

The heterogeneity of opinion in the literature on the impact of radiotherapy makes patient information and decision-making difficult. It may be that the detrimental effect of radiotherapy is outweighed in terms of patient satisfaction by the benefit of immediate reconstruction with a definitive reconstruction and that surgeons' concerns are overvalued, yet it is upon this anecdotal surgeon-reported outcome that patient decision making is based.

In an era when breast cancer patients are more likely to survive their disease (85% for 5 year survival), the physical and psychological effects of treatment, especially long term effects, are very relevant. A woman with residual dissatisfaction with her reconstructed breast has a constant reminder of her disease and treatment. Optimising reconstructive outcomes is a major issue in survivorship.

Rationale

Surgeons strive to attain the best possible reconstructive outcomes and are aware of the effects of radiotherapy on an autologous flap. They therefore often advise against any procedure which may have a detrimental impact on "their" flap. However, from a patient perspective, by having a delayed reconstruction the treatment pathway is prolonged by several months, if not years, and requires an additional operation(s) compared to those who undergo immediate reconstruction and PMRT. There remains significant uncertainty in the literature about the magnitude of the impact of radiotherapy from a surgeon's perspective and very little is known about the patients' preferences in terms of detrimental impact on flap vs effect of the prolonged pathway on their lives.

By objectively assessing irradiated autologous flap reconstructions and comparing with unirradiated patients we will understand further the impact of radiotherapy on an autologous flap. By quantifying the difference in patient satisfaction, and understanding the perspective of patients who have PMRT to an immediate or delayed reconstruction we will understand further the impact of both pathways on their lives, the reconstruction and their satisfaction with the result. This, we believe, will enable clinicians to better inform patients, empowering them in their decision-making about the best timing for breast reconstruction and potentially enabling more women to undergo immediate definitive breast reconstruction with DIEP flap.

We intend to enrol patients who have undergone unilateral mastectomy and DIEP reconstruction. Patients will fall into one of four possible groups depending on the decision made by the surgeon and patient pre-operatively.

Patient groups:

1. Unilateral skin sparing mastectomy (SSM) with immediate DIEP flap reconstruction and PMRT (cases)
2. Unilateral SSM with immediate DIEP flap reconstruction and no PMRT (controls)
3. Unilateral simple mastectomy, PMRT, and subsequent delayed DIEP flap reconstruction (controls)
4. Unilateral SSM with temporizing implant, PMRT and subsequent conversion to DIEP (controls)

The study will be conducted as a mixed methods case control study using both quantitative and qualitative research methods. Initially a prospective study was planned, however for those patients who undergo a delayed reconstruction the whole oncological and reconstructive process can take several years. Secondly the number of patients who are currently undergoing radiotherapy to their DIEP breast reconstruction is relatively small. For these reasons it was decided that a truly prospective study would not be practical but prospective data collection from a recent cohort of patients would yield a greater study population.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have undergone one of the treatment sequences above (a) - (d)

   Patient groups:
   1. Unilateral skin sparing mastectomy (SSM) with immediate DIEP flap reconstruction and PMRT (cases)
   2. Unilateral SSM with immediate DIEP flap reconstruction and no PMRT (controls)
   3. Unilateral simple mastectomy, PMRT, and subsequent delayed DIEP flap reconstruction (controls)
   4. Unilateral SSM with temporizing implant, PMRT and subsequent conversion to DIEP (controls)
2. Patients of any age will be included
3. Patients who are between one and five years post initial breast reconstruction surgery or radiotherapy (which ever is most recent)

Exclusion Criteria:

1. Women who have undergone bilateral mastectomy, even if the contralateral mastectomy was asynchronous.
2. Women who are less than one year from their last radiotherapy treatment or from their DIEP flap reconstruction.
3. Patients who have had more than one implant based operation before DIEP flap (revision surgery to the implant implies that an implant based reconstruction was the primary intent and therefore the DIEP flap is a 'salvage' procedure) or if it is documented to be a salvage reconstruction.
4. Women who have developed recurrent / distant disease.
5. Women who are unable to stand for the 3D imaging (approximately 10 minutes)
6. Women who are unable to complete the English language questionnaire or interview (i.e. learning difficulties or patients who do not have adequate English language skills).

   -

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who has undergone unilateral DIEP reconstruction for breast cancer at the Royal Marsden NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01-14; Primary Completion 2018-01-14 (Estimated); Study Completion 2018-01-14 (Estimated)

PRIMARY OUTCOMES:
The difference in patient satisfaction score between patients with an irradiated DIEP flap (group (a)) and patients with a DIEP flap who have not undergone PMRT (group (b)) using "satisfaction with reconstructed breast" question of the BREAST-Q. | Day 1
  The difference in (mean or median) patient satisfaction score (ranging from 0-100) between patients with an irradiated DIEP flap (group (a)) and patients with a DIEP flap who have not undergone PMRT (group (b)) using the "satisfaction with reconstructed breast" subscale of the postoperative reconstruction module of the BREAST-Q questionnaire.

SECONDARY OUTCOMES:
The difference in scores in other subscales from the BREAST-Q questionnaire between patients with an irradiated DIEP flap (group (a)) and patients with a DIEP flap who have not undergone PMRT (group (b)). | Day 1
The difference in patient satisfaction and all subscales between patients with an irradiated DIEP flap (group (a)) and patients who underwent PMRT prior to DIEP flap (group (c) and group (d)) using BREAST-Q scores as above. | Day 1
Volume and symmetry assessment of the reconstructed breast using 3D surface imaging This would consist of comparing volume and symmetry assessment between groups (a) and (b), groups (a) and (c), and groups (a) and (d). | Day 1
Panel assessment by independent panel of the reconstruction using 3D surface imaging. | Day 1
  The panel will consist of four members, a plastic surgeon, a breast surgeon, a clinical oncologist and a breast care nurse. The panel will score independently. The scoring will be between 1 and 4
Applanation tonometry for assessment of the consistency of the reconstructed breast. This will consist of comparing breast compressibility in the reconstructed breast between groups (a) and (b), groups (a) and (c), and groups (a) and (d). | Day 1
The prevalence of fat necrosis. | Day 1
  The presence of fat necrosis would be either:
  Presence of fat necrosis (as documented by imaging) - Yes or no Surgical procedure (excluding biopsy) to treat fat necrosis - Yes or no This would consist of comparing prevalence of fat necrosis and surgical procedures required. Rates of each would be compared between groups (a) and (b), groups (a) and (c), and groups (a) and (d).
The number of operative episodes for the index breast and the contralateral breast. | Day 1
  One visit to theatre counts as one operative episode (i.e. if multiple procedures to the same breast on one occasion then this is still just one operative episode).
  This would consist of comparing number of episodes in the index breast and the contra lateral breast between groups (a) and (b), groups (a) and (c), and groups (a) and (d).
Analysis of time from diagnosis to definitive breast reconstruction or last radiotherapy session This would consist of a comparison of number of months treatment between group (a) and group (c), group (a) and group (d). | Day1
Knowledge of patient experience from interviews regarding patient satisfaction. Please refer to methodology for further details. | Day 1
Basic health economics of the four treatment groups. This will include cost of each operation/inpatient episodes for all breast related operations and cost of all plastic surgical outpatient events. | Day 1
Median length of time between end of treatment to time of the study for each of the groups a to d. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rusby, DM FRCS, Principal Investigator — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Derived] O'Connell RL, Di Micco R, Khabra K, Kirby AM, Harris PA, James SE, Power K, Ramsey KWD, Rusby JE. Comparison of Immediate versus Delayed DIEP Flap Reconstruction in Women Who Require Postmastectomy Radiotherapy. Plast Reconstr Surg. 2018 Sep;142(3):594-605. doi: 10.1097/PRS.0000000000004676. PMID 29927832